CLINICAL TRIAL: NCT03282812
Title: Cancer Prevention Study-II Nutrition Cohort
Brief Title: Metabolomics and Breast Cancer Risk in a Nested Case-control Study of the Cancer Prevention Study-II Nutrition Cohort
Status: Completed | Type: Observational
Sponsor: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: CPSII_BRCA_NCC
Record Dates: First submitted 2017-09-11; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases
- controls

SUMMARY:
This study aims to investigate diet, lifestyles, serum metabolomics in relation to breast cancer risk in a nested case-control study including 1,547 postmenopausal women from the Cancer Prevention Study II (CPS-II) Nutrition Cohort. The CPS-II Nutrition Cohort is a prospective cohort study of cancer incidence and mortality among 184,185 men and women, established by the American Cancer Society in 1992. Participants completed a self-administered baseline questionnaire in 1992/1993 including demographic, medical, and lifestyle information. Follow-up questionnaires were sent to living participants in 1997 and every other year to update exposure information and ascertain newly diagnosed cancers. From June 1998 through May 2001, blood specimens were collected from 21,963 women. All participants completed a short questionnaire and provided informed consent at the time of blood draw. Non-fasting whole blood collected from each participant was shipped chilled overnight to a central repository, processed, and frozen in liquid nitrogen at approximately -130 °C for long-term storage.

Of the 21,963 women who provided a blood sample, investigators identified 782 postmenopausal women diagnosed with invasive breast cancer between blood draw date and June 2011 who had not been diagnosed with cancer (other than nonmelanoma skin cancer) before blood draw or prior to their breast cancer diagnosis. Controls were 1:1 matched to cases on date of birth, date of blood draw, and race and were cancer free at the date of case diagnosis. Seventeen women who were selected as controls were later diagnosed with breast cancer, at which time they became a case. A total of 1,547 postmenopausal women were included in the breast cancer nested case-control study.

ELIGIBILITY:
Inclusion Criteria:

* blood sample
* cancer free at blood draw

Exclusion Criteria:

* unverified breast cancer
* non-invasive breast cancer

Min Age: 50 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1547 (Actual)
Dates: Start 1998-06 (Actual); Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Incident invasive breast cancer | Blood draw through June 30, 2011
  Identified through medical record or linkage with state cancer registry

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Calle EE, Rodriguez C, Jacobs EJ, Almon ML, Chao A, McCullough ML, Feigelson HS, Thun MJ. The American Cancer Society Cancer Prevention Study II Nutrition Cohort: rationale, study design, and baseline characteristics. Cancer. 2002 May 1;94(9):2490-501. doi: 10.1002/cncr.101970. PMID 12015775
- [Derived] Wang Y, Gapstur SM, Carter BD, Hartman TJ, Stevens VL, Gaudet MM, McCullough ML. Untargeted Metabolomics Identifies Novel Potential Biomarkers of Habitual Food Intake in a Cross-Sectional Study of Postmenopausal Women. J Nutr. 2018 Jun 1;148(6):932-943. doi: 10.1093/jn/nxy027. PMID 29767735